CLINICAL TRIAL: NCT06935396
Title: Comparison of Muscle Strength, Functional Exercise Capacity, Physical Activity Level, and Quality of Life Between Insulin-Using and Non-Insulin-Using Patients With Type 2 Diabetes
Brief Title: Comparison of Physical Function and Quality of Life in Insulin and Non-Insulin Users With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Ayşen Karaman, MSc. PT., Eastern Mediterranean University
Other Study IDs: DAU-2025-T2D-INS01
Record Dates: First submitted 2025-04-17; First posted 2025-04-20 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; muscle strength; quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Insulin-Using Type 2 Diabetes: Participants in this group are Type 2 Diabetes patients who are using insulin therapy. No specific drug dosage is administered as part of this study; the group is simply observed based on their existing insulin treatment regimen.
- Non-Insulin-Using Type 2 Diabetes: This group consists of patients diagnosed with Type 2 Diabetes who are not using insulin. They may be managing their condition through oral medications or lifestyle changes, but no specific intervention is provided within the scope of this study.
- Healthy Controls: This group consists of healthy individuals with no history of Type 2 Diabetes or any other chronic conditions. No medical intervention or treatment is administered, and they serve as a control group for comparison with the diabetic groups.

SUMMARY:
This clinical trial aims to compare the muscle strength, functional exercise capacity, physical activity levels, and quality of life between insulin-using and non-insulin-using patients with Type 2 diabetes. The study will involve participants aged 40-70, diagnosed with Type 2 diabetes, and will assess their physical performance through a series of standardized tests. The primary objective is to determine if insulin use impacts the physical fitness and overall health of patients with Type 2 diabetes. Results from this study could lead to better management strategies for diabetic patients.

DETAILED DESCRIPTION:
This study aims to analyzemuscle strength, functional exercise capacity, physical activity levels, and quality of life (QoL) among a control group, insulin-using, and non-insulin-using patients with Type 2 Diabetes Mellitus. A total of 67 individuals with a mean age of 54.68 ± 7.41 years were included in the study. Among these participants, 18 were insulin users (Group 1), 21 were non-insulin users (Group 2) with Type II Diabetes, and 28 were healthy individuals (Group 3). Demographic data of the participants were recorded. Grip strength was measured using a hand-grip dynamometer, and quadriceps strength was measured with a handheld dynamometer. Functional exercise capacity was evaluated using the 6-minute walk test (6 MWT), and physical activity levels were assessed using the International Physical Activity Questionnaire (IPAQ). The Short Form-12 questionnaire was used to assess QoL, the 30-second sit-to-stand test was used for lower extremity strength, and the Semmes-Weinstein Monofilament test was conducted to evaluate protective sensory loss.

ELIGIBILITY:
Inclusion Criteria:

* Must have been diagnosed with Type 2 Diabetes Mellitus by a specialist doctor at least 5 years ago
* Must be between 40-65 years of age
* Must have signed the informed consent form
* Must be literate

Exclusion Criteria:

* Presence of active diabetic foot ulcer
* History of acute trauma affecting the musculoskeletal system within the last month
* Presence of musculoskeletal, orthopedic, neurological, or cardiopulmonary diseases
* Participants who are unable to cooperate to the extent that they cannot understand the given instructions

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals diagnosed with Type 2 Diabetes Mellitus (T2DM). Participants will be divided into three groups:
  Insulin-using T2DM patients.
  Non-insulin-using T2DM patients.
  Healthy controls (no history of diabetes or chronic diseases).
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Grip Strength | This measurement was taken once at the time of study participation to evaluate the baseline strength level in all groups.
  Grip strength was measured using a hand-held dynamometer, where participants squeezed the device with maximal force to record the strength
Functional Exercise Capacity | This measurement was taken once at baseline
  Functional exercise capacity was assessed using the 6-minute walk test (6MWT). Participants walked as far as possible in 6 minutes, and the total distance walked was recorded
Quality of Life SF-12 | Measurement was taken once at baseline
  Quality of life was assessed using the Short Form-12 (SF-12) questionnaire. This questionnaire evaluates general health, physical functioning, and mental well-being. It consists of 12 questions selected from the Short Form - 36 (SF-36) quality of life questionnaire. The SF-12 includes the following subcomponents: physical functioning, physical role, pain, general health, emotional role, mental health, social functioning, and vitality.
  A Physical Component Summary Score (PCS), which represents the physical domain of quality of life, was calculated from the subcomponents of physical functioning, physical role, general health, and pain.
  A Mental Component Summary Score (MCS) was calculated from the subcomponents of emotional role, mental health, vitality, and social functioning.
  Each subcomponent and summary score ranges from 0 to 100, with higher scores indicating better quality of life.
Lower Extremity Strength | Measurement was taken once at baseline
  Lower extremity strength was assessed using the 30-second sit-and-stand test. Participants were asked to rise from a seated position and sit back down repeatedly within 30 seconds, and the total number of repetitions was recorded.
Protective Sensory Loss | Measurement was taken once at baseline
  rotective sensory loss was assessed using the Semmes-Weinstein Monofilament Test. This test is used to assess the sensation of touch in the feet, particularly for loss of protective sensation.
Physical Activity Level | Measurement was taken once at baseline
  Physical activity level was assessed using the International Physical Activity Questionnaire (IPAQ).The International Physical Activity Questionnaire Short Form (IPAQ-SF) will be used to determine the level of physical activity. The Turkish validity and reliability study has been conducted, and the test-retest reliability was found to be r = 0.69. This form is self-administered and consists of seven questions covering the "last seven days" to assess the level of physical activity. It provides information about the time spent sitting, walking, and engaging in moderate- and vigorous-intensity activities. A score is calculated by multiplying the minutes, days, and MET value. For the calculation, a MET value of 8 is used for vigorous physical activity, 4 for moderate-intensity activity, and 3.3 for walking. Since the scale is open access, it does not require permission for use (

CONTACTS AND LOCATIONS:
Overall Officials: Ayşen Karaman, MSc, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Mersin, Famagusta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It has not yet been determined whether individual participant data (IPD) will be shared.